CLINICAL TRIAL: NCT03801538
Title: The Optimizing Treatment of Peginterferon Alpha in Chronic Hepatitis B Patients With Low Level HBsAg(I-Cure-3X)
Brief Title: The Optimizing Treatment of Peginterferon Alpha in Chronic Hepatitis B Patients With Low Level HBsAg
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Zhiliang Gao, Professor, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I-Cure-3X
Record Dates: First submitted 2019-01-09; First posted 2019-01-11 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Nucleosides; nas

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PEG-IFN group (Experimental): patients were treated with NAs once a day and PEG-IFN once a week for 12 weeks. At week 12, the decrease of HBsAg was evaluated.
  ①If the decrease of HBsAg is more than 50%. NAs was stopped. PEG-IFN Treatment was continued for a prolonged period (no more than 96 weeks) until the endpoint was achieved, or terminated in week 96.
  ②If the decrease of HBsAg is less than 50%.NAs and PEG-IFN was extended to week 24. Then, If the decrease of HBsAg is more than 50%. NAs was stopped, PEG-IFN Treatment was continued for a prolonged period (no more than 96 weeks) until the endpoint was achieved, or terminated in week 96. If the decrease of HBsAg is less than 50%. PEG-IFN was stopped, patients were treated with NAs once a day and then followed up for 48 weeks.
  Interventions: Drug: Peginterferon Alfa
- NAs group (Other): CHB patients do not need to change their NAs treatment.
  Interventions: Drug: Nucleoside Analog (Substance)

INTERVENTIONS:
Drug: Peginterferon Alfa — Peginterferon Alfa-2A 180 micrograms/week or Peginterferon Alfa-2B 180 micrograms/week, for at most 96 weeks.
  Other Names: PEG-IFN
  Arms: PEG-IFN group
Drug: Nucleoside Analog (Substance) — Patients do not need to change their NAs treatment.
  Other Names: NAs
  Arms: NAs group

SUMMARY:
HBeAg-negative chronic hepatitis B (CHB) patients with low Level HBsAg were enrolled. After giving informed consent, patients were treated with nucleoside analog(s) (NAs) once a day and weekly subcutaneous injections of peginterferon alfa-2a 180 micrograms/week or peginterferon alfa-2b 180 micrograms/week for 12 weeks. At week 12, the decrease of HBsAg was evaluated.

①If the decrease of HBsAg is more than 50% compared to baseline level. NAs was stopped, patients were treated with weekly subcutaneous injections of alfa-2a 180 micrograms/week or peginterferon alfa-2b 180 micrograms/week. Treatment endpoint was HBsAg loss(<0.05 IU/ mL). Depending on the decline of HBsAg level, treatment was either continued for a prolonged period (no more than 96 weeks) until the endpoint was achieved, or terminated in week 96. After treatment, all patients were followed up for 48 weeks.

②If the decrease of HBsAg is less than 50% compared to baseline level. The combination therapy of NAs and peginterferon alfa was extended to week 24. Then, the decrease of HBsAg was evaluated again.

If the decrease of HBsAg is more than 50% compared to baseline level. NAs was stopped, patients were treated with weekly subcutaneous injections of alfa-2a 180 micrograms/week or peginterferon alfa-2b 180 micrograms/week. Treatment endpoint was HBsAg loss(<0.05 IU/mL). Depending on the decline of HBsAg level, treatment was either continued for a prolonged period (no more than 96 weeks) until the endpoint was achieved, or terminated in week 96. After treatment, all patients were followed up for 48 weeks.

If the decrease of HBsAg is less than 50% compared to baseline level. Peginterferon alfa was stopped, patients were treated with NAs once a day and then followed up for 48 weeks.

Patients who maintained the original NAs treatment served as a control group.

DETAILED DESCRIPTION:
It is estimated that more than 400 million people are infected with hepatitis B virus (HBV) globally. HBeAg-negative CHB patients with low Level HBsAg were enrolled in the out-patient department of Third Affiliated Hospital of Sun Yat-sen University and Wuhan Union Hospital. All of them were HBsAg positive and anti-HBs negative for more than 6 months with HBV DNA<100 IU/mL and HBsAg levels <1000 IU/mL. All patients did not have other liver diseases and contraindications for interferon therapy. After giving informed consent, patients were treated with nucleoside analog(s) (NAs) once a day and weekly subcutaneous injections of peginterferon alfa-2a 180 micrograms/week or peginterferon alfa-2b 180 micrograms/week for 12 weeks. At week 12, the decrease of HBsAg was evaluated.

①If the decrease of HBsAg is more than 50% compared to baseline level. NAs was stopped, patients were treated with weekly subcutaneous injections of alfa-2a 180 micrograms/week or peginterferon alfa-2b 180 micrograms/week. Treatment endpoint was HBsAg loss(<0.05 IU/ mL). Depending on the decline of HBsAg level, treatment was either continued for a prolonged period (no more than 96 weeks) until the endpoint was achieved, or terminated in week 96. After treatment, all patients were followed up for 48 weeks.

②If the decrease of HBsAg is less than 50% compared to baseline level. The combination therapy of NAs and peginterferon alfa was extended to week 24. Then, the decrease of HBsAg was evaluated again.

If the decrease of HBsAg is more than 50% compared to baseline level. NAs was stopped, patients were treated with weekly subcutaneous injections of alfa-2a 180 micrograms/week or peginterferon alfa-2b 180 micrograms/week. Treatment endpoint was HBsAg loss(<0.05 IU/mL). Depending on the decline of HBsAg level, treatment was either continued for a prolonged period (no more than 96 weeks) until the endpoint was achieved, or terminated in week 96. After treatment, all patients were followed up for 48 weeks.

If the decrease of HBsAg is less than 50% compared to baseline level. Peginterferon alfa was stopped, patients were treated with NAs once a day and then followed up for 48 weeks.

The use of other immune suppressive or regulatory drugs and other antiviral drugs was prohibited during the course of the study. In this study, HBsAg loss(<0.05 IU/mL) was defined as treatment endpoint. Anti-HBs positive(>10 milli-International unit)(mIU/mL) was defined as seroconversion.

Patients who maintained the original NAs treatment served as a control group.

ELIGIBILITY:
Inclusion Criteria:

1. CHB patients who had received NAs for more than 12 months.
2. Hepatitis B e antigen (HBeAg)-negative.
3. Hepatitis B surface antigen (HBsAg) positive and <1000 IU/mL.
4. Hepatitis B virus DNA <100 IU/mL.

Exclusion Criteria:

1. Patients with liver cirrhosis, Hepatocellular Carcinoma or alpha feto protein (AFP) >2 upper limit of normal(ULN) or other malignancies.
2. Patients with other factors causing liver diseases.
3. Pregnant and lactating women.
4. Patients with concomitant HIV infection or congenital immune deficiency diseases.
5. Patients with diabetes, autoimmune diseases.
6. Patients with important organ dysfunctions.
7. Patients with serious complications (e.g., infection, hepatic encephalopathy, hepatorenal syndrome, gastrointestinal bleeding.)
8. Patients who receive antineoplastic or immunomodulatory therapy in the past 12 months.
9. Patients who can't come back to clinic for follow-up on schedule.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
HBsAg Clearance | 96 weeks
  Participants with HBsAg <0.05 IU/mL.
HBsAg Seroconversion | 96 weeks
  Participants with HBsAg <0.05 IU/mL and anti-HBsAg positive

CONTACTS AND LOCATIONS:
Overall Officials: Zhiliang Gao, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- Department of Infectious Diseases, The Third Affliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided